CLINICAL TRIAL: NCT00482027
Title: A Phase 1 Randomized, Placebo-controlled, Double-blind Dose-escalation Trial to Evaluate the Safety and Immunogenicity of tgAAC09, a Gag-PR-RT AAV HIV Vaccine
Brief Title: Safety and Immunogenicity Study of tgAAC09, a Gag-PR-RT AAV HIV Vaccine
Acronym: A001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Targeted Genetics Corporation (Industry); Children's Hospital of Philadelphia (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: A001
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2007-05

CONDITIONS: HIV Infection
Keywords: HIV vaccine; Adeno-associated virus vactored vaccine; HIV-1 subtype C; Safety; Immunogenicity; Biodistribution; HIV prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 AAV-2 HIV Vaccine (Active Comparator): 64 volunteers receiving AAV-2 HIV vaccine tgAAC09 at 3 dosage levels, dose escalation and dose optimization
  Interventions: Biological: tgAAC09
- 2 (Placebo Comparator): 16 volunteers receiving formulation buffer consisting of a buffered salt solution with potassium phosphate, calcium chloride, magnesium chloride, and HEPES

INTERVENTIONS:
Biological: tgAAC09 — one or 2 doses of AAV-2 HIV vaccine (tgAAC09) at 3 dosage levels, dose escalation and dose optimization
  Other Names: AAV-2 HIV Vaccine
  Arms: 1 AAV-2 HIV Vaccine

SUMMARY:
The purpose of this study is to determine safety and immunogenicity (ability to induce an immune response) of a novel HIV vaccine based on adeno-associated virus (AAV)

DETAILED DESCRIPTION:
The need for a vaccine to prevent AIDS and interrupt transmission of HIV is indisputable. To be effective, an HIV vaccine will have to induce cellular and humoral immune responses that are durable and potent. Intra-muscular delivery of HIV genes enclosed within recombinant adeno-associated virus (rAAV) protein capsid has been shown to be a potent inducer of both antibodies and T-cell responses in animal studies. tgAAC09, consisting of single-stranded DNA from Clade C HIV-1 genes for the gag, protease and part of the reverse transcriptase proteins enclosed within a rAAV serotype 2 protein capsid, was developed as one component of a multi-component HIV vaccine. The purpose of this study is to evaluate the safety and immunogenicity of tgAAC09 in healthy, HIV-seronegative volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age at least 18 years on the day of screening and no greater than 50 years on the day of vaccination
* Available for follow-up for the planned duration of the study (screening plus 12 months)
* Able to give written informed consent;
* No reported high-risk behavior for HIV (Appendix C), willing to undergo HIV testing and receive results;
* If sexually active, willing to use or have partner use condoms from screening until at least 4 months after the vaccination. Additional means of contraception are permitted and encouraged.

Exclusion Criteria:

* Clinically relevant abnormality on history or examination including history of immunodeficiency or use of immunosuppressive medication in last 6 months;
* A chronic medical condition or concurrent condition, which, in the opinion of the investigator, would make the volunteer unsuitable for the study.
* Any of the following abnormal laboratory parameters that are mild and judged to be clinically significant by the principal investigator or designee, or moderate, severe, or very severe: hematology (hemoglobin, absolute neutrophil count [ANC] absolute lymphocyte count [ALC], absolute CD4 count, platelets); urinalysis, clinical chemistry (total bilirubin, creatinine, AST, ALT). Refer to Appendix D for the grading of these laboratory parameters.
* If female, pregnant or planning a pregnancy within 4 months after receiving the vaccine, or lactating;
* Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of vaccination;
* Receipt of other experimental HIV vaccine at any time;
* Receipt of blood transfusion or blood products within 6 months of vaccination;
* Participation in another clinical trial of an investigational product currently or within 12 weeks of vaccination, or expected during participation in this study;
* History of severe local or systemic reaction to vaccination or history of allergic reactions to vaccines;
* Confirmed infection with HIV-1 or HIV-2;
* Positive for hepatitis B (surface antigen), hepatitis C antibodies, or active syphilis (confirmed by treponemal test such as TPHA in addition to non-treponemal test such as RPR) or active tuberculosis.
* Unlikely to comply with protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety of one or two doses of tgAAC09 | One year
  Safety of one or two doses of tgAAC09 at 3 dosage levels in a dose-escalating an ddose-optimization study

SECONDARY OUTCOMES:
Immunogenicity | up to 6 months post 2nd injection

OTHER OUTCOMES:
Biodistribution | upt to 6 montsh post 1st injection

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mehendale, MD, Principal Investigator — National AIDS Research Institute; Nathan Clumeck, MD, Principal Investigator — St. Pierre University Hospital; Jan van Lunzen, MD, Principal Investigator — University of Hamburg-Eppendorf
Locations (5):
- Belgium (2):
  - SGS Biopharma, Antwerp
  - St. Pierre University Hospital, Brussels
- Germany (2):
  - Univeristy of Bonn, Bonn
  - University of Hamburg, Hamburg
- National AIDS Research Institute, Pune, India

REFERENCES:
- [Result] Mehendale S, van Lunzen J, Clumeck N, Rockstroh J, Vets E, Johnson PR, Anklesaria P, Barin B, Boaz M, Kochhar S, Lehrman J, Schmidt C, Peeters M, Schwarze-Zander C, Kabamba K, Glaunsinger T, Sahay S, Thakar M, Paranjape R, Gilmour J, Excler JL, Fast P, Heald AE. A phase 1 study to evaluate the safety and immunogenicity of a recombinant HIV type 1 subtype C adeno-associated virus vaccine. AIDS Res Hum Retroviruses. 2008 Jun;24(6):873-80. doi: 10.1089/aid.2007.0292. PMID 18544020
- [Derived] Vardas E, Kaleebu P, Bekker LG, Hoosen A, Chomba E, Johnson PR, Anklesaria P, Birungi J, Barin B, Boaz M, Cox J, Lehrman J, Stevens G, Gilmour J, Tarragona T, Hayes P, Lowenbein S, Kizito E, Fast P, Heald AE, Schmidt C. A phase 2 study to evaluate the safety and immunogenicity of a recombinant HIV type 1 vaccine based on adeno-associated virus. AIDS Res Hum Retroviruses. 2010 Aug;26(8):933-42. doi: 10.1089/aid.2009.0242. PMID 20666584